CLINICAL TRIAL: NCT04087434
Title: HOAC: Improving Health Outcomes for Acute Concussion Patients
Brief Title: Health Outcomes for Acute Concussion
Acronym: HOAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kendra Jorgensen-Wagers (U.S. Federal Agency)
Collaborators: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kendra Jorgensen-Wagers, Senior Clinical Research Director, Office of Naval Research (ONR)
Organization: Office of Naval Research (ONR) (U.S. Federal Agency)
Other Study IDs: N00014-18-C-2019
Record Dates: First submitted 2019-04-23; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Brain Injury, Acute
Keywords: concussion
MeSH Terms: conditions — Brain Injuries; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective: retrospective review of 300 records of patients following concussive diagnosis to track recovery and adherence to progressive return to activity recommendations.
- Prospective: 300 prospective patients enrolled following concussive diagnosis to track recovery, clinical diagnosis and brain gauge performance.
  Interventions: Device: Brain Gauge Prospective and Healthy Control
- Control Group: 75-100 Healthy Controls recruited by Fort Bragg to assess performance in a healthy population for brain gauge performance.
  Interventions: Device: Brain Gauge Prospective and Healthy Control

INTERVENTIONS:
Device: Brain Gauge Prospective and Healthy Control — The Brain Gauge is a brain health assessment system that takes advantage of the well-documented relationship between the sensory nerves in the fingers and the projection of those nerves to corresponding regions in the brain. The system is composed of a test device (the Brain Gauge) that uses novel fingertip vibration patterns to probe cortical complexity and utilize that complexity to gain more sensitive and specific detection of compromised neural function.
  Groups: Control Group; Prospective

SUMMARY:
The primary purpose of this prospective observational trial is to validate the Brain Gauge device as an objective tool for concussion assessment and treatment in order to determine if a method that has proven successful in 18-22 year old collegiate student-athletes will be applicable for military personnel. Overall aims of the study include:

1. Demonstration that the Brain Gauge can objectively measure concussion in this population and thus improve concussion identification and coding.
2. Demonstration of stronger screening for and tracking of acute concussion and documentation of concussion diagnoses, including improved tracking of recovery and greater adherence to DOD/VA Clinical Practice Guidelines for acute concussion.

DETAILED DESCRIPTION:
The primary purpose of this prospective observational trial is to validate the Brain Gauge device as an objective tool for concussion assessment and treatment in order to determine if a method that has proven successful in 18-22 year old collegiate student-athletes will be applicable for military personnel. Overall aims of the study include: Demonstration that the Brain Gauge can objectively measure concussion in this population and thus improve concussion identification and coding; Demonstration of stronger screening for and tracking of acute concussion and documentation of concussion diagnoses, including improved tracking of recovery and greater adherence to DOD/VA Clinical Practice Guidelines for acute concussion.

A retrospective cohort of 300 anonymized patients from Landstuhl Regional Medical Center will be used as historical controls to assess diagnosis and recovery patterns, while a comparison cohort of 100 healthy active duty members from Fort Bragg, NC, will be used as uninjured controls to establish baseline Brain Gauge metrics in this population.

For the prospective cohort, all participants will receive comprehensive standard of care medical assessment and treatment as determined by their clinical team and as appropriate to their injury and course of recovery. In addition to standard assessments, participants will complete the Brain Gauge assessments at home or in the clinic at selected time points from initial assessment through 90 days post-study entry. The Brain Gauge system is designed for use by the patient at home and is easily incorporated in a remote, tele-health based patient monitoring system.

Data will be analyzed for compliance with current military Clinical Practice Guidelines (CPGs) for mTBI, both with the use of the Brain Gauge system and prior to its implementation. Objective cortical neurofunctional measures from the Brain Gauge instrument will be compared to standardized clinical measures.

ELIGIBILITY:
Inclusion Criteria

* Active duty military aged 18-60 stationed within local catchment area.
* Confirmed concussion within the last 72 hours

Exclusion Criteria

* a sensory, motor or central neurological disorder such as seizures, ADD/ADHD, autism or neuropathy in the hands.
* Subtest test records incomplete for key variables such as symptom report inventories.
* Current MEB in process.
* Pregnant women as there are parts of the Clinical practice guide that cannot be implemented as a part of standard clinical care due to pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Active duty service members with or without a concussion diagnosis within the past 7 days.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-01-10 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Validate Brain Gauge to detect clinical/ statistically significant change in reaction time, reaction time variability, temporal order judgment, accuracy,fatigue and stimulus discrimination between concussed and healthy controls.. | 90 days
  The Brain Gauge is a health assessment system that takes advantage of the relationship between the sensory nerves in the fingers and the projection of those nerves to the corresponding regions in the brain. The system is composed of a mouse sized test device that uses novel fingertip vibration patterns to probe cortical connectivity and utilize that connectivity to gain more sensitive and specific detection of neural function. In sports concussion studies using this technology has established efficacy for detecting mild traumatic brain injury and tracking its recovery for differentiating individuals with and without traumatic brain injury with no baseline measures required.

SECONDARY OUTCOMES:
Examine utility of remote telehealth clinical oversight for TBI recovery to improve accountability, and responsibilities for tracking concussion recovery | over the course of a year
  Prove efficacy of assessment via remote capability with synchronous and asynchronous Telehealth clinical oversight from TBI trained staff. This trial utilizes a symptom tracking application that patients can deploy on their own phones and complete the neurobehavioral symptom inventory. Mild traumatic brain injuries are difficult to diagnose or assess and are particularly difficult to assess in circumstances were triage decisions are necessary. Use of the Brain Gauge device as well as a patient centered commercial off the shelf software is hypothesized to not only increase patient compliance in treatment but also significantly personalize treatment to foster stronger recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Kendra L Jorgensen-Wagers, Ph.D, Principal Investigator — The Defense and Veterans Brain Injury Center
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No